CLINICAL TRIAL: NCT05334862
Title: Residual Torsional Deformity in Pediatric Genu Varum After Coronal Plane Deformity Correction by 8 Plate Hemi Epiphysiodesis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Nasseh Hafeez Boles, Resident doctor, Orthopaedic surgery department, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8 plate in genu varum
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Paediatric Surgery

STUDY DESIGN:
Intervention Model Description: skeletally immature patients over 2.5 years of age and less than 12 years of age who presented with genu varum. (unilateral or bilateral)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- skeletally immature patients between 2.5 : 12 years with genu varum (Active Comparator): skeletally immature patients over 2.5 years of age and less than 12 years of age who presented with genu varum. (unilateral or bilateral) ..those will be treated by 8 plate hemi epiphysiodesis.
  Interventions: Procedure: 8 plate hemiepiphysiodesis

INTERVENTIONS:
Procedure: 8 plate hemiepiphysiodesis — surgical procedure by lateral incision in proximal tibia and distal femur and fixation by using 8 plate and screws.

SUMMARY:
This study is to evaluate the residual torsional deformity in pediatric Genu Varum after coronal plane deformity correction by 8 plate hemi epiphysiodesis.

DETAILED DESCRIPTION:
Angular deformities around the knee in children is a common finding including genu valgum and genu varum.

The genu valgum or varum may be idiopathic or arise from diverse etiologies, such as trauma, dysplasia, metabolic disease, inflammatory, endocrine, tumor, neoplastic, or developmental pathologies.

Surgical treatment options include osteotomies with either acute or gradual correction and temporary hemi epiphysiodesis (guided growth),the latter being less invasive and with significantly lower rate of major complications.

Guided growth by 8 plate hemi epiphysiodesis is commonly used to correct coronal plane deformity around the knee. Since its introduction by Stevens in 2007 many studies have demonstrated the efficacy, safety and advantages of tension band plating in the paediatric age group as an alternative to corrective osteotomy.

Genu varum deformities of the leg are often associated with internal tibial torsion. The 3 major causes of pediatric in-toeing are metatarsus adductus, internal tibial torsion, and femoral anteversion.

..yet, there is no enough available literature studies evaluating the amount of correction of torsional deformity after coronal plane deformity correction by 8 plate hemi epiphysiodesis.

This is the question of this study and we are trying to answer it by measuring the residual torsional deformity after achieving full correction of coronal plane deformity by 8 plate hemi epiphysiodesis.

ELIGIBILITY:
- Inclusion criteria: skeletally immature patients over 2.5 years of age and less than 12 years of age who presented with genu varum. (unilateral or bilateral)

- Exclusion criteria:

1. skeletal maturity.
2. epiphyseal dysplasia.
3. metabolic and neurologic disorders.
4. previous trauma.
5. patients younger than 2.5 years and older than 12 years old

Ages: 30 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
residual torsional deformity measured via clinical examination. | 1 year
  clinical examination by measuring : thigh foot angle - foot progression angle - heel bisector - internal and external rotaion of the hip

SECONDARY OUTCOMES:
Any complications detected | 1 year
  Follow up of the patient postoperatively and clinical examination. Number of participants with any complications

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elbaseet, Doctor, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from october 2025
Access Criteria: anyone

REFERENCES:
- [Background] Schleien CL, Eberle B, Shaffner DH, Koehler RC, Traystman RJ. Reduced blood-brain barrier permeability after cardiac arrest by conjugated superoxide dismutase and catalase in piglets. Stroke. 1994 Sep;25(9):1830-4; discussion 1834-5. doi: 10.1161/01.str.25.9.1830. PMID 8073465
- [Background] Parzuchowski A, Winiarska K. [Cataract surgery in patients with pronounced disorders of general condition]. Klin Oczna. 1972;42(4):1032-7. No abstract available. Polish. PMID 5072935